CLINICAL TRIAL: NCT05720689
Title: Contribution of Music During Dental Care Under MEOPA in Children
Brief Title: Music During Dental Children Care Under MEOPA
Acronym: SONOMEOPAeDENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20-API-03
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Dental Diseases
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison by cross-over
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEOPA dental care with music (Experimental): diffusion of relaxing music during dental care under MEOPA
  Interventions: Other: using relaxing music
- MEOPA dental care without music (Active Comparator): dental care under MEOPA as usual
  Interventions: Other: No relaxing music

INTERVENTIONS:
Other: using relaxing music — music diffusion during dental care under MEOPA
  Arms: MEOPA dental care with music
Other: No relaxing music — dental care under MEOPA without music
  Arms: MEOPA dental care without music

SUMMARY:
In France, the improvement of dental care for children in general and even more so for children with special needs is a real public health issue. Indeed, children under 6 years of age, children with a fear that is difficult to control and who have failed to receive care, or children with disabilities, have difficulties in receiving care. Because of their medical wandering before effective therapeutic care, they are up to 4 times more likely to have a very degraded oral health condition involving avulsions rather than conservative care. Moreover, these complex situations often lead to the indication of dental care under conscious sedation with an equimolar mixture of oxygen and nitrous oxide (MEOPA) or even under general anesthesia (GA); hospital sedation by administration of midazolam is exceptionally proposed. As access to GA care is largely insufficient, solutions likely to improve the success rate of care and anxiolysis provided by MEOPA associated with cognitive-behavioral management must be considered.

Among these, music has been shown to have variable neurophysiological effects (action on cardiac and respiratory rhythms and on blood pressure), depending on the style of music used. During dental care, a biological and psychological impact on emotion has been highlighted, although the few studies carried out in children in this particular context are not at a high level of proof. In children with special needs, the addition of music to MEOPA could therefore increase relaxation or distraction during dental care and improve the success rate of sedation by MEOPA. Validation of this hypothesis would limit the redirection of the young patient under GA and prevent the loss of opportunity associated with a further delay in care of several months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 12 years referred for dental care under sedation in one of the four HU dental services
* Children requiring at least two sessions of the same type and duration
* Consent of the holders of parental authority, consent of the children
* Health coverage for the child (social security affiliation)
* Child and parents are French speaking and able to communicate with the medical team

Exclusion Criteria:

* Contraindications to the use of MEOPA
* Nasal breathing disorders such as a flu syndrome ("blocked nose" not allowing nasal ventilation)
* Hearing impaired children
* Patients with complications during inhalation (especially headaches)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Success of sedation (binary) according to the Venham scale modified by Veerkamp | 1 day
  (success: scores 0-1-2; failure: scores 3-4-5)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Lille University hospital, Lille
  - Marseille University hospital, Marseille
  - Nice University Hospital, Nice
  - Toulouse University hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No